CLINICAL TRIAL: NCT05876546
Title: Assessment of the Primary, Accumulated Irritability and Skin Sensitization Potential of an Elastic Collodion-based Liquid Bandage Under Controlled and Maximized Conditions (RIPT)
Brief Title: Evaluation of Skin Irritancy and Sensitization of a Liquid Bandage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: EF184A
Record Dates: First submitted 2023-04-27; First posted 2023-05-25 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-02

CONDITIONS: Skin Care
Keywords: Contact test; HRIPT
MeSH Terms: interventions — Abortion, Induced

STUDY DESIGN:
Intervention Model Description: Induction period (3 weeks): the experimental and control product will be applied through a patch test on the participants' back for 3 consecutive weeks, with 3 weekly applications, with the first week being the primary irritation phase and the two consecutive weeks being the irritation phase. accumulated irritation. Rest period (10 to 15 days): corresponds to the rest period, when participants will remain without any contact test applied to their back, which will follow the induction period, where there will be no application of the experimental and control product. Challenge period (3 days): the experimental and control product will be applied to the participants' back, in a naïve area. Products will be removed after 48 hours, with readings taking place after removal and approximately 24 hours after removal. This period corresponds to the sensitization phase.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liquid bandage (Experimental): liquid bandage - The liquid bandage will be distributed on a contact test filter paper disc, appropriately identified, in the letter of the alphabet corresponding to the experimental product.
  Interventions: Device: Liquid bandage
- Saline Solution (Sham Comparator): saline solution - The sterile saline solution (NaCl 0.9%) will be used as control in another contact test filter paper disc, appropriately identified, in the letter of the alphabet corresponding to the control.
  Interventions: Device: Saline Solution

INTERVENTIONS:
Device: Liquid bandage — The liquid bandage will be applied through a patch test to the participants' backs for 3 consecutive weeks, with 3 weekly applications. Afterwards, there will be a rest period of between 10 and 15 days. The liquid bandage will be applied again to the participants' back, in a naive area and removed after 48 hours.
  Arms: Liquid bandage
Device: Saline Solution — The saline solution will be applied via patch test to the participants' backs for 3 consecutive weeks, with 3 weekly applications. Afterwards, there will be a rest period of between 10 and 15 days. The saline solution will be applied again to the participants' back, in a naive area and removed after 48 hours.
  Arms: Saline Solution

SUMMARY:
The investigational product constitutes a medical device that is freely accessible to consumers and, as such, must be safe under real or reasonably foreseeable conditions of use and its safety must be tested before being placed on the market.

Therefore, this study was designed to evaluate the biocompatibility of the experimental product, as provided for in legislation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old.
* Fitzpatrick phototype I to IV.
* Presence of intact skin in the test region.
* Agreement to comply with the study procedures and requirements and attend the institute on the days and times determined for the assessments.
* Signature of the Informed Consent Form (ICF) before carrying out any study procedure.

Exclusion Criteria:

* Presence of skin marks in the test region that interfere with the assessment of possible skin reactions (for example, pigmentation disorders, vascular malformations, scars, increased hairiness, large quantities of ephelides and nevus, sunburn).
* Presence of active dermatosis (local or disseminated) that could interfere with the study results.

istory of atopy (atopic dermatitis, allergic rhinitis, allergic bronchitis, allergic conjunctivitis, etc.).

- History of allergic reactions, irritation or intense sensations of discomfort to topical products such as, for example, cosmetics, health products or medicines.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Prove the absence of primary irritability potential of the experimental product under maximized conditions. | 6 weeks
  * Occurrence of primary irritation;
  * Occurrence of accumulated irritation;
  * Occurrence of sensitization;
  * Occurrence of AEs ;
  * Treatment discontinuations due to AEs . It is expected that after the study period, the product will be considered safe because it does not promote a positive irritability response and skin sensitization in the study group. No statistical inference analysis will be performed. The results will be presented in the form of tables demonstrating whether or not there was a positive response of irritability or skin sensitization in the study group. During the study, the regions of the product and control application will be evaluated and if any clinical sign is found, it will be classified according to the scale recommended by the International Contact Dermatitis Research Group - ICDRG - (FISHER, 1995).

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Allergisa, Campinas, São Paulo
  - Eurofarma Laboratorios S.A, São Paulo